CLINICAL TRIAL: NCT05609071
Title: Technology of Intracranial Pressure Estimation by Single-Channel EEG in Brain Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SNUEMSBDICP
Record Dates: First submitted 2022-10-30; First posted 2022-11-08 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Intracranial Pressure Increase; Brain Diseases
Keywords: Electroencephalogram; Intensive care unit; Intracranial pressure monitoring
MeSH Terms: conditions — Intracranial Hypertension; Brain Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
If intracranial pressure can be measured non-invasively using single-channel EEG, clinicians will be able to easily monitor changes in intracranial pressure in patients with brain diseases in the clinical setting. Therefore, a more efficient treatment plan can be established and the prognosis of patients with brain disease can be expected to improve in the long term.

DETAILED DESCRIPTION:
Study Objectives:

1. Accuracy evaluation of single-channel EEG-based estimated intracranial pressure and actual intracranial pressure in patients with brain disease
2. It is intended to improve the accuracy by analyzing and upgrading the correlation and concordance of the single-channel EEG-based estimated intracranial pressure compared with the actual intracranial pressure measurement of the patient.

Study design: Multi-center prospective clinical trial

The study procedure was explained to the caregiver of the patient with brain disease admitted to the emergency room or intensive care unit, who was or will be implanted with an intracranial pressure monitoring device and informed consent was obtained.

While the intracranial pressure monitoring device is being applied, EEG data and intracranial pressure data are simultaneously acquired by applying a single-channel EEG.

EEG-based intracranial pressure prediction model and actual intracranial pressure comparison analysis are conducted to evaluate the prediction model and upgrade it.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patients have had or are planning to insert an intracranial pressure monitoring device due to brain diseases
* Emergency room or intensive care unit of the study hospital

Exclusion Criteria:

* EEG measurement is restricted due to trauma or head deformity
* The attachment of electrodes for EEG measurement interferes with the standard treatment
* Patients who do not agree to enroll to this study by patients or caregivers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is intended for patients admitted to the intensive care unit (ICU) who are adults (18 years or older) and who are undergoing intracranial pressure measurement for some type of brain disease. Except for cases where the 2-channel EEG cannot be attached, it is intended for patients who can acquire EEG.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference between estimated intracranial pressure and actual intracranial pressure | through study completion, an average of 1 year
  The difference between the estimated intracranial pressure and the actual intracranial pressure is calculated using the previously developed intracranial pressure prediction formula using quantitative EEG parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Ki Hong Kim, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University HOspital, Seoul, South Korea